CLINICAL TRIAL: NCT06950489
Title: A Feasibility Study of Tegoprazan and Amoxicillin Dual Therapy for the Treatment of Helicobacter Pylori
Brief Title: Tegoprazan and Amoxicillin Dual Therapy
Status: Recruiting | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2025
Record Dates: First submitted 2025-04-28; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: H.Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dual therapy for Helicobacter pylori refers to a treatment regimen that combines two agents: a potent acid suppressor (such as a proton pump inhibitor [PPI] or a potassium-competitive acid blocker [PCAB]) and the antibiotic amoxicillin. This approach is increasingly recognized as a viable alternative to traditional triple or quadruple therapies, particularly in the context of rising resistance to other antibiotics such as clarithromycin and metronidazole. Potent acid suppression increases the stability and activity of amoxicillin against H. pylori by maintaining a higher gastric pH, which is essential for optimal amoxicillin effect. High-dose dual therapy (e.g., amoxicillin 1,000 mg three times daily + standard dose of PPI three or four times daily for 14 days) has demonstrated eradication rates of 90%. In 2015, vonoprazan, a novel P-CAB, was launched in Japan and used as an alternative for PPIs for eradicating H. pylori. Dual therapy with vonoprazan and amoxicillin is particularly effective, with cure rates comparable to triple therapy and superior outcomes in clarithromycin-resistant infections. Dual therapy is generally well tolerated, with adverse event rates similar to or lower than those seen with triple or quadruple regimens. In 2018, a new P-CAB, tegoprazan, was developed in Korea and approved for H. pylori eradication. However, there was no study of tegoprazan and amoxicillin dual therapy for the treatment of H. pylori.

DETAILED DESCRIPTION:
The investigators aim to evaluate the H. pylori eradication success rate and treatment compliance of tegoprazan and amoxicillin dual therapy.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* Drug allergy to antibiotics
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rates | 6 weeks
  Urea breath test after completing H. pylori eradication regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea